CLINICAL TRIAL: NCT01163981
Title: A Randomised Controlled Trial of the Effectiveness of Ultrasound Guidance in Cannulation of Dialysis Arteriovenous Fistulas and Grafts in a University Hospital Dialysis Unit
Brief Title: Ultrasound Guided Cannulation of Dialysis Fistulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Access 5
Record Dates: First submitted 2010-07-12; First posted 2010-07-16 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2018-10

CONDITIONS: Haemodialysis
Keywords: duplex Ultrasound; Haemodialysis; Vascular Access
MeSH Terms: interventions — Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blind cannulation (No Intervention): Cannulation without guidance
- Ultrasound guided cannulation (Experimental): Ultrasound guided cannulation
  Interventions: Other: Use of ultrasound guidance in cannulation

INTERVENTIONS:
Other: Use of ultrasound guidance in cannulation — Use of guidance with duplex ultrasound to complete cannulation of dialysis access
  Other Names: duplex ultrasound
  Arms: Ultrasound guided cannulation

SUMMARY:
The investigators suspect that using ultrasound to guide insertion of needles for dialysis patients will make this process quicker and more accurate, thus reducing complications and reducing discomfort for patients.

DETAILED DESCRIPTION:
Haemodialysis patients need to have two needles inserted into a large surgically altered vein (fistula) or surgical vascular graft/shunt for every dialysis session. Some fistulas or shunts may be more difficult to insert needles into than others. As such a system of colour coding or "traffic lighting" of patients is in place in most units. A "green light" patient is easy to "needle" with two needles and the majority of staff within the unit will be able to connect the patients to the dialysis machine. A "red light" patient is reserved for the more experienced staff within the unit who will often have to be timetabled to work specific times so that they are present to connect certain patients to the dialysis machines. "Amber light" fistulas lie between these two extremes.

Ultrasound (US) is routinely used in many hospitals and many dialysis units will have access to a machine to assess patients for problems. Indeed central venous line insertions for dialysis are now almost always performed under US guidance since two large studies in this area in 2002 provided strong evidence that US guided placement significantly reduces complications during catheter placement and a reduction in the number of attempts at insertion. In addition the National Institute of Clinical Excellence in the UK provided evidence that insertion time is quicker although this association was statistically less convincing.

Ultrasound offers the advantage of dynamic imaging without the risks of radiation exposure and can be done as an office based procedure using portable equipment.

Studies in emergency departments and particularly in paediatric care have suggested that US guidance can improve the speed and accuracy of cannulation in peripheral veins for intravenous access.

We suggest that US guided cannulation of fistulas might improve the cannulation rate of more difficult fistulas and potentially reduce the time required to commence dialysis and the number of local complications of cannulation (haematoma/aneurysm/infection).

To our knowledge US is not used in cannulation guidance in any dialysis units, although most units will have access to a machine as above. We therefore propose to perform a randomised controlled trial of US guided cannulation of fistulas versus current practice (blind cannulation) to assess the effectiveness of US controlled cannulation in a busy dialysis unit.

ELIGIBILITY:
Inclusion criteria:

1. Dialysis 3X per week
2. Dialysing via 2 needles in fistula
3. No deviation from routine dialysis protocol (additional or no heparin etc)

Exclusion criteria:

a. Active or recent fistula infection/thrombosis/intervention in 6/52 of study

Withdrawal criteria:

1. Patient request
2. Patient non compliance with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Time to establish dialysis | Within an average of 5 minutes into each of the next 12 consecutive dialysis session
  Time to commence 2 needle dialysis from first palpation or imaging of fistula

SECONDARY OUTCOMES:
- Patient reported pain scores Patient reported anxiety and pain | enrollment, two weeks and four weeks into trial
  Patient reported pain scores and anxiety scores recorded by questionnaire
Number of cannulation attempts( skin punctures or passes of needle) | Within an average of 5 minutes into each of the next 12 consecutive dialysis session
  number of cannulation attempts required
complications of needling | Within 2 hours of completing each of the next 12 consecutive dialysis sessions
  record presence of any complications due to needle insertion
Referral for difficult needling during trial | From enrollment to 24 hours following completion of the last of 12 consecutive dialysis sessions
  Referral for difficult needling to either senior nurse or to access clinic during trial

CONTACTS AND LOCATIONS:
Overall Officials: George E Smith, BSc MBBS MRCS, Principal Investigator — Hull and East Yorkshire NHS Trust
Locations (1):
- Hull Royal Infirmary, Hull, East Yorkshire, United Kingdom